CLINICAL TRIAL: NCT05361252
Title: Restrictive Versus Liberal Stroke Volume Variation-guided Fluid Infusion in Major Liver Tumour Resection: a Prospective Randomised Trial of Perioperative Quality of Care
Brief Title: Stroke Volume Variation-guided Fluid Infusion in Major Liver Tumour Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yuan-Yi Chia, Chief of Anesthesiology, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS16-CT8-25
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Fluid Management
Keywords: Stroke volume variation; Fluid therapy; Hepatectomy; Alanine aminotransferase; Estimated glomerular filtration rate

STUDY DESIGN:
Intervention Model Description: This trial had a randomised study design with simple randomisation and a fixed allocation ratio (1:1 to the low-SVV group or high-SVV group). The patients were blinded to the randomisation and allocation.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the low-SVV group (Active Comparator): the value of stroke volume variation will be less than or equal to 10 this group
  Interventions: Procedure: SVV-guided fluid management
- the high-SVV group (Active Comparator): the value of stroke volume variation will be higher than 10 this group
  Interventions: Procedure: SVV-guided fluid management

INTERVENTIONS:
Procedure: SVV-guided fluid management — fluid will be guided by value of stroke volume variation

SUMMARY:
Studies have demonstrated that the rate of change in stroke volume variation (SVV) can be used to determine the volume of body fluids during major abdominal surgery. Anaesthesiologists can use SVV as a guide for the appropriate administration of intraoperative fluids to improve postoperative prognoses. Liver surgery is a major abdominal operation, and the amount of blood lost is typically higher than that during other general abdominal surgeries. Blood loss is positively correlated with the intraoperative fluid infusion volume, and greater blood loss is associated with more postoperative complications. Additionally, comorbid liver disease or cirrhosis can increase the complexity of liver tumour resection, causing difficulty in assessing intravascular volume and determining the appropriate intraoperative infusion volume.

ELIGIBILITY:
Inclusion Criteria:

* We initially selected 118 patients who required hepatectomy.
* The physiological status of the patients was assessed in terms of American Society of Anesthesiologists scores I-III

Exclusion Criteria:

* Extreme body mass index (BMI)
* Age under 20 or over 75 years
* Emergency surgery
* Preexisting cardiac, hepatic, renal, or coagulation disorder; hyperthyroidism; and sinus arrhythmia.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative complications in the two groups. | From day 1 to day 30 after surgery.
  calculate the incidence of postoperative complication within 30 days

SECONDARY OUTCOMES:
The differences of perioperative ALT | Examination report on the 1st postoperative day.
  Calculate the difference of the perioperative physiological variables
The differences of perioperative eGFR | Examination report on the 1st postoperative day.
  Calculate the difference of the perioperative physiological variables
The differences of perioperative creatinine | Examination report on the 1st postoperative day.
  Calculate the difference of the perioperative physiological variables
The differences of perioperative T.bil | Examination report on the 1st postoperative day.
  Calculate the difference of the perioperative physiological variables
The differences of perioperative Hb | Examination report on the 1st postoperative day.
  Calculate the difference of the perioperative physiological variables
The differences of perioperative arterial lactate | Examination report on the 1st postoperative day.
  Calculate the difference of the perioperative physiological variables
The differences of perioperative albumin | Examination report on the 1st postoperative day.
  Calculate the difference of the perioperative physiological variables
The pain scale | up to three days postoperatively
  Assessment of postoperative pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Yi Chia, Director, Principal Investigator — Kaohsiung Veterans General Hospital.; Kai-Wei Hsieh, physician, Study Director — Kaohsiung Veterans General Hospital.; We-Yu Chen, physician, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang K, Boldt J, Suttner S, Haisch G. Colloids versus crystalloids and tissue oxygen tension in patients undergoing major abdominal surgery. Anesth Analg. 2001 Aug;93(2):405-9 , 3rd contents page. doi: 10.1097/00000539-200108000-00034. PMID 11473870 (Retraction: PMID 21451066 Anesth Analg. 2011 May;112(5):1211)
- [Background] Mythen MG, Webb AR. The role of gut mucosal hypoperfusion in the pathogenesis of post-operative organ dysfunction. Intensive Care Med. 1994;20(3):203-9. doi: 10.1007/BF01704701. No abstract available. PMID 8014287
- [Background] Sear JW. Kidney dysfunction in the postoperative period. Br J Anaesth. 2005 Jul;95(1):20-32. doi: 10.1093/bja/aei018. Epub 2004 Nov 5. PMID 15531622
- [Background] Osman D, Ridel C, Ray P, Monnet X, Anguel N, Richard C, Teboul JL. Cardiac filling pressures are not appropriate to predict hemodynamic response to volume challenge. Crit Care Med. 2007 Jan;35(1):64-8. doi: 10.1097/01.CCM.0000249851.94101.4F. PMID 17080001
- [Background] Tavernier B, Makhotine O, Lebuffe G, Dupont J, Scherpereel P. Systolic pressure variation as a guide to fluid therapy in patients with sepsis-induced hypotension. Anesthesiology. 1998 Dec;89(6):1313-21. doi: 10.1097/00000542-199812000-00007. PMID 9856704
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Su NY, Huang CJ, Tsai P, Hsu YW, Hung YC, Cheng CR. Cardiac output measurement during cardiac surgery: esophageal Doppler versus pulmonary artery catheter. Acta Anaesthesiol Sin. 2002 Sep;40(3):127-33. PMID 12434609
- [Background] Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, Fleming SC. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. Br J Anaesth. 2005 Nov;95(5):634-42. doi: 10.1093/bja/aei223. Epub 2005 Sep 9. PMID 16155038
- [Background] Lefrant JY, Bruelle P, Aya AG, Saissi G, Dauzat M, de La Coussaye JE, Eledjam JJ. Training is required to improve the reliability of esophageal Doppler to measure cardiac output in critically ill patients. Intensive Care Med. 1998 Apr;24(4):347-52. doi: 10.1007/s001340050578. PMID 9609413
- [Background] Lopes MR, Oliveira MA, Pereira VO, Lemos IP, Auler JO Jr, Michard F. Goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery: a pilot randomized controlled trial. Crit Care. 2007;11(5):R100. doi: 10.1186/cc6117. PMID 17822565
- [Background] McKendry M, McGloin H, Saberi D, Caudwell L, Brady AR, Singer M. Randomised controlled trial assessing the impact of a nurse delivered, flow monitored protocol for optimisation of circulatory status after cardiac surgery. BMJ. 2004 Jul 31;329(7460):258. doi: 10.1136/bmj.38156.767118.7C. Epub 2004 Jul 8. PMID 15242867
- [Background] Boldt J, Ince C. The impact of fluid therapy on microcirculation and tissue oxygenation in hypovolemic patients: a review. Intensive Care Med. 2010 Aug;36(8):1299-308. doi: 10.1007/s00134-010-1912-7. Epub 2010 May 26. PMID 20502873 (Retraction: PMID 32405741 Intensive Care Med. 2020 Jun;46(6):1301)
- [Background] Rahbari NN, Zimmermann JB, Schmidt T, Koch M, Weigand MA, Weitz J. Meta-analysis of standard, restrictive and supplemental fluid administration in colorectal surgery. Br J Surg. 2009 Apr;96(4):331-41. doi: 10.1002/bjs.6552. PMID 19283742
- [Background] Choi JM, Lee YK, Yoo H, Lee S, Kim HY, Kim YK. Relationship between Stroke Volume Variation and Blood Transfusion during Liver Transplantation. Int J Med Sci. 2016 Feb 20;13(3):235-9. doi: 10.7150/ijms.14188. eCollection 2016. PMID 26941584
- [Background] Correa-Gallego C, Tan KS, Arslan-Carlon V, Gonen M, Denis SC, Langdon-Embry L, Grant F, Kingham TP, DeMatteo RP, Allen PJ, D'Angelica MI, Jarnagin WR, Fischer M. Goal-Directed Fluid Therapy Using Stroke Volume Variation for Resuscitation after Low Central Venous Pressure-Assisted Liver Resection: A Randomized Clinical Trial. J Am Coll Surg. 2015 Aug;221(2):591-601. doi: 10.1016/j.jamcollsurg.2015.03.050. Epub 2015 Apr 7. PMID 26206652
- [Background] Lim C, Audureau E, Salloum C, Levesque E, Lahat E, Merle JC, Compagnon P, Dhonneur G, Feray C, Azoulay D. Acute kidney injury following hepatectomy for hepatocellular carcinoma: incidence, risk factors and prognostic value. HPB (Oxford). 2016 Jun;18(6):540-8. doi: 10.1016/j.hpb.2016.04.004. Epub 2016 May 7. PMID 27317959
- [Background] Slankamenac K, Breitenstein S, Held U, Beck-Schimmer B, Puhan MA, Clavien PA. Development and validation of a prediction score for postoperative acute renal failure following liver resection. Ann Surg. 2009 Nov;250(5):720-8. doi: 10.1097/SLA.0b013e3181bdd840. PMID 19809295
- [Background] Saner F. Kidney failure following liver resection. Transplant Proc. 2008 May;40(4):1221-4. doi: 10.1016/j.transproceed.2008.03.068. PMID 18555153
- [Background] Peres LA, Bredt LC, Cipriani RF. Acute renal injury after partial hepatectomy. World J Hepatol. 2016 Jul 28;8(21):891-901. doi: 10.4254/wjh.v8.i21.891. PMID 27478539
- [Background] Jarnagin WR, Gonen M, Fong Y, DeMatteo RP, Ben-Porat L, Little S, Corvera C, Weber S, Blumgart LH. Improvement in perioperative outcome after hepatic resection: analysis of 1,803 consecutive cases over the past decade. Ann Surg. 2002 Oct;236(4):397-406; discussion 406-7. doi: 10.1097/01.SLA.0000029003.66466.B3. PMID 12368667
- [Background] Moug SJ, Smith D, Wilson IS, Leen E, Horgan PG. The renal sequelae of a novel triphasic approach to blood loss reduction during hepatic resection. Eur J Surg Oncol. 2006 May;32(4):435-8. doi: 10.1016/j.ejso.2006.01.011. Epub 2006 Mar 7. PMID 16520017
- [Background] Giannini EG, Testa R, Savarino V. Liver enzyme alteration: a guide for clinicians. CMAJ. 2005 Feb 1;172(3):367-79. doi: 10.1503/cmaj.1040752. PMID 15684121
- [Background] Olthof PB, Huiskens J, Schulte NR, Wicherts DA, Besselink MG, Busch OR, Heger M, van Gulik TM. Postoperative peak transaminases correlate with morbidity and mortality after liver resection. HPB (Oxford). 2016 Nov;18(11):915-921. doi: 10.1016/j.hpb.2016.07.016. Epub 2016 Sep 2. PMID 27600437
- [Background] Siu J, McCall J, Connor S. Systematic review of pathophysiological changes following hepatic resection. HPB (Oxford). 2014 May;16(5):407-21. doi: 10.1111/hpb.12164. Epub 2013 Aug 29. PMID 23991862
- [Background] Yu LH, Yu WL, Zhao T, Wu MC, Fu XH, Zhang YJ. Post-operative delayed elevation of ALT correlates with early death in patients with HBV-related hepatocellular carcinoma and Post-hepatectomy Liver Failure. HPB (Oxford). 2018 Apr;20(4):321-326. doi: 10.1016/j.hpb.2017.10.001. Epub 2018 Jan 17. PMID 29373299
- [Background] Choi SS, Kim SH, Kim YK. Fluid management in living donor hepatectomy: Recent issues and perspectives. World J Gastroenterol. 2015 Dec 7;21(45):12757-66. doi: 10.3748/wjg.v21.i45.12757. PMID 26668500